CLINICAL TRIAL: NCT07377084
Title: Metabolomics of Cancers of the Upper Aerodigestive Tract
Acronym: METABORL
Status: Recruiting | Type: Observational
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Other Study IDs: 2020/14
Record Dates: First submitted 2025-02-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Upper AerodigestiveTract Cancer
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with upper aerodigestive tract tumor requiring a panendoscopy with biopsy
  Interventions: Procedure: Blood samples for the analysis of sildenafil in plasma; Biological: urine samples

INTERVENTIONS:
Procedure: Blood samples for the analysis of sildenafil in plasma — blood samples collection at screening and between the 3rd and 6th month after the end of treatment.
Biological: urine samples — Urine samples collection at screening and between the 3rd and 6th month after the end of treatment.

SUMMARY:
Metabolomics, thanks to advances in mass spectrometry, allows for the analysis of cellular metabolites to better understand biological processes. In oncology, it provides a global view of metabolic alterations in tumors and enables the classification of cancers based on various medical parameters using advanced statistical methods (machine learning). Its low cost and speed make it a promising approach in personalized medicine.

Cancers of the upper aerodigestive tract (UADT), the fifth most common cancer in France, are often diagnosed late, reducing survival chances (35-50% at five years). Identifying a specific metabolomic signature for these cancers could facilitate early detection, assess treatment response, and rapidly detect recurrences. Additionally, HPV-induced tumors may exhibit a distinct metabolic profile compared to those caused by tobacco and alcohol. Currently, no published studies have explored this topic for UADT cancers, highlighting the need for such research.

The aim of this study is to identify a metabolomic signature associated with the presence of UADT cancer at initial diagnosis and during post-therapeutic follow-up (three months after treatment completion). Hypothesis is that a specific metabolomic signature will be observed in the biological samples of patients diagnosed with UADT cancer, that the type of observed signature could be correlated with tumor site, stage, HPV status, and prognosis, and that the persistence or disappearance of this metabolomic signature three months after treatment may be associated with the risk of recurrence. The search for this potential metabolomic signature will be conducted using tumor biopsies, plasma, and urine samples at the initial diagnostic phase and plasma and urine samples at three and six months post-treatment follow-up.

Ultimately, the benefits of this study lie in improving early diagnosis, treatment (adjusting treatment based on the prognostic value of specific metabolomic signatures), and follow-up (early detection of recurrences, adapting monitoring to each patient's individual risk) of UADT cancers.

As the study is based on biological samples collected as part of standard patient care (with no additional biological tests or procedures performed specifically for research), no research-related risk is expected for the patient.

This is a prospective, single-center study involving patients with histologically confirmed, untreated squamous cell carcinoma of the UADT (oral cavity, oropharynx, larynx, and hypopharynx) who will receive curative treatment at the Antoine Lacassagne Center.

The search for a potential metabolomic signature will be conducted using biological and tumor samples collected as part of standard patient care, without requiring additional tests or procedures.

The primary objective of the study is to identify a metabolomic signature in patients with UADT cancer.

The secondary objectives of the study are:

* To investigate the correlation between a metabolomic signature and tumor characteristics.
* To examine the relationship between a metabolomic signature at three to six months post-treatment and oncological status at three to six months and one year post-treatment in patients with UADT cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven squamous cell carcinoma of the upper aerodigestive tract (oral cavity, oropharynx, larynx, and hypopharynx), stage T1-4, N0-3, M0, untreated.
* Curative treatment planned at CAL.
* Patient who has voluntarily consented to the use of their data and signed a non-opposition form for the use of their biological and tumor samples.

Exclusion Criteria:

* Metastatic patient (M1).
* No curative treatment possible.
* History of cancer (other than basal cell carcinoma) in the last 5 years.
* Tumor size deemed insufficient according to the assessment of the ENT surgeon.
* Patient refusal to allow the use of their biological and tumor samples for research.
* Vulnerable persons are defined in articles L1121-5 to -8:

  * Pregnant women, women in labor, and nursing mothers, individuals deprived of liberty by a judicial or administrative decision, individuals hospitalized without consent under articles L. 3212-1 and L. 3213-1 who are not covered by the provisions of article L. 1121-8,
  * And individuals admitted to a health or social establishment for purposes other than research,
  * Adults under legal protection or unable to express their non-opposition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes patients managed for a suspected upper aerodigestive tract tumor undergoing ENT panendoscopy with biopsies, with final inclusion limited to patients with histologically confirmed squamous cell carcinoma of the upper aerodigestive tract.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-11-04 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure is the diagnostic performance (sensitivity/specificity) of the metabolomic signature in patients with UADT cancer. | At screening and between the 3rd and 6th month after the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre BOZEC, MD, Principal Investigator — Centre Antoine Lacassagne
Locations (1):
- Centre Antoine Lacassagne, Nice, France